CLINICAL TRIAL: NCT01812083
Title: Interleukin-1 Receptor Antagonist Gene Polymorphism and Adverse Pregnancy Outcome in Turkish Women
Acronym: IRAGPAAOITW
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Nilgün Özlem Alptekin, Dental Faculty, Selcuk University
Other Study IDs: SelcukU; SUDHF1451 (Registry Identifier: SUDHF1451)
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Periodontitis
Keywords: Periodontitis; adverse pregnancy outcomes; IL-1 polymorphism
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators hypothesized that the IL-1A (+4895), IL-1B (+3954), and IL-1RN gene polymorphisms may be associated with PLBW. Smoking has been well documented by numerous studies as a major environmental risk factor for periodontitis and adverse pregnancy outcomes. Therefore, the investigators only selected non-smoking individuals in this study as the smoking-related risk could obscure the polymorphism-related increase in risk for periodontitis and adverse pregnancy outcomes. This study aimed to determine the association between IL-1A (+4895), IL-1B (+3954), and IL-1RN polymorphisms with adverse pregnancy outcomes and periodontitis in a non-smoking Turkish population.

DETAILED DESCRIPTION:
Pregnant women between 18-35 years of age with single gestation and with ≥20 on-crowded teeth excluding third molars were included in this study. Subjects were divided into normal birth (NB) and PLBW groups on the basis of their pregnancy outcome. Women who delivered an infant with a birth weight of more than 2500 g after 37 weeks of gestation were placed in the NB group. Women who delivered infants whose birth weight was below 2500 g or before 37 weeks of gestation were placed in the PLBW group. Current/past tobacco user, alcohol abuse, history of high-risk gestation, hypertension, gestational diabetes, any systemic disease and placenta previa were the exclusion criteria for this study. Maternal, obstetric, and demographic factors such as maternal age, maternal education, regular prenatal care, genitourinary tract infections during pregnancy, total number of births, previous PLBW, and antibiotic use during the pregnancy period were also recorded.

ELIGIBILITY:
Inclusion Criteria:

Subjects were divided into normal birth (NB) and PLBW groups on the basis of their pregnancy outcome. Women who delivered an infant with a birth weight of more than 2500 g after 37 weeks of gestation were placed in the NB group.

Exclusion Criteria:

Current/past tobacco user, alcohol abuse, history of high-risk gestation, hypertension, gestational diabetes, any systemic disease and placenta previa were the exclusion criteria for this study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women between 18-35 years of age with single gestation and with ≥20 on-crowded teeth excluding third molars were included in this study. Subjects were divided into normal birth (NB) and PLBW groups on the basis of their pregnancy outcome. Women who delivered an infant with a birth weight of more than 2500 g after 37 weeks of gestation were placed in the NB group. Women who delivered infants whose birth weight was below 2500 g or before 37 weeks of gestation were placed in the PLBW group.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2004-01; Primary Completion 2004-06 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Interleukin-1 receptor antagonist gene polymorphism and adverse pregnancy outcome in Turkish women | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Özlem Alptekin, DDS,PhD,Prof, Study Chair — Selcuk University Faculty of Dentistry